CLINICAL TRIAL: NCT01244646
Title: Perceived Hypoglycemia- and Weight-related Quality of Life of Patients With Sulfonylurea Derivate-treated Diabetes Mellitus Type 2, a Non-interventional Study.
Brief Title: Hypoglycemia- and Weight-related Quality of Life in Patients With Diabetes Mellitus Type 2 on Sulfonylurea Derivatives.
Status: Terminated | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CNL-DUM-2010/1
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus; Type 2; DMT2; T2DM; metformin; sulfonylurea; hypoglycemia; weight; quality of life; compliance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypoglycemia; Body Weight; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Diabetes Mellitus Type 2

SUMMARY:
1. A prospective, non-interventional study, 125 patients with Diabetes Mellitus Type2 will be enrolled, who, while on metformin, have a sub-optimal glycemic control and who thus will receive additional treatment with a sulfonylurea (SU) derivative. At the start and at 3 and 6 months, during regular visits to the patient's General Practitioner, the patients will complete a series of questionnaires (Patient Reported Outcomes, PROs) directed at diabetes in general, at fear for hypoglycemia, at body weight, at treatment compliance and at general wellbeing. These PROs are the worry subscale of the Hypoglycaemic Fear Survey, Impact of Weight on Quality of Life, revised Diabetes Symptom Checklist, Problem Areas In Diabetes, EuroQol EQ-5D and Medication Adherence Report Scale. In total 75 questions. The frequency of hypoglycemic symptoms, incidence of hypoglycemic events and body weight changes will be assessed and the level of adherence to treatment will be investigated.
2. Diabetic patients, M/F, aged >35, metformin treated, serum HbA1c ≥7.0% (within last month), informed consent provided, in whom a SU therapy is added. Patients with Type 1 diabetes and with secondary diabetes will be excluded, and patients unable to understand and complete the questionnaires.
3. Primary outcome variables are outcomes from HFS-w and IWQOL in relation to the frequency of hypoglycemic symptoms and body weight at 6 months and to weight change from 0 to 6 months. Secondary outcome variables are the other PROs. The frequency of hypoglycemic symptoms, incidence of hypoglycemic events, changes in body weight and level of compliance will be addressed.
4. The Intention To Treat analysis will be used, with Last Value Extended Forward from 3 to 6 months in case of withdrawal after 3 months. Changes in outcome variables will be analysed by modelling time and potential dummy variables in a Generalized Estimating Equations analysis.
5. Secondary, outcomes in HFS-w and IWQOL are compared with self-reported hypoglycemic symptoms, incidence of hypoglycemic events, body weight and change in body weight from 0 to 6 months. Changes in all PRO's from 0 to 3 and 6 months, potential relationships between (changes in) the different questionnaires, such as with hypoglycemia symptoms, weight (changes) and treatment compliance will be evaluated. A search is done for baseline characteristics which predict outcomes and changes in PRO's, hypoglycemic symptoms, hypoglycemic events and weight changes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus Type 2 for > 6 months on treatment with only metformin for >4 weeks
* HbA1c value >7.0 and therefore a sulfonylurea derivative is added
* Able to complete a series of questionnaires

Exclusion Criteria:

* Concomitant treatment with an other antidiabetic than metformin and SU derivative
* Contraindications for the use of metformin or SU derivative
* Concomitant diseases which may affect the patient's ability to complete study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General practitioners, group practices in primary care, pharmacists
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Hypoglycemic Fear Survey (HFS) questionnaire | 0 months
Hypoglycemic Fear Survey (HFS) questionnaire | 3 months
Hypoglycemic Fear Survey (HFS) questionnaire | 6 months
Impact of Weight on Quality of Life (IWQOL-Lite) questionnaire | 0 months
Impact of Weight on Quality of Life (IWQOL-Lite) questionnaire | 3 months
Impact of Weight on Quality of Life (IWQOL-Lite) questionnaire | 6 months

SECONDARY OUTCOMES:
Diabetes Symptom Checklist (DSC-R) questionnaire, | 0 months
Diabetes Symptom Checklist (DSC-R) questionnaire, | 3 months
Diabetes Symptom Checklist (DSC-R) questionnaire, | 6 months
Medication Adherence Report Scale (MARS-5) questionnaire | 0 months
Medication Adherence Report Scale (MARS-5) questionnaire | 3 months
Medication Adherence Report Scale (MARS-5) questionnaire | 6 months
Investigator-asked Symptoms of Hypoglycemia, hypoglycemic events, weight, compliance | 0 months
Investigator-asked Symptoms of Hypoglycemia, hypoglycemic events, weight, compliance | 3 months
Investigator-asked Symptoms of Hypoglycemia, hypoglycemic events, weight, compliance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. F.J. Snoek, PhD, Study Chair — VU University of Amsterdam
Locations (22):
- Netherlands (22):
  - Research Site, Alkmaar
  - Research Site, Edam
  - Research Site, Gorinchem
  - Research Site, Heerhugowaard
  - Research Site, Heiloo
  - Research Site, Hoogvliet
  - Research Site, Lichtenvoorde
  - Research Site, Limmen
  - Research Site, Maasbracht
  - Research Site, Noord-Scharwoude
  - Research Site, Poortvliet
  - Research Site, Rotterdam
  - Research Site, Spijkenisse
  - Research Site, The Hague
  - Research Site, Tuitjenhorn
  - Research Site, Vaassen
  - Research Site, Valkenswaard
  - Research Site, Voerendaal
  - Research Site, Volendam
  - Research Site, Wamel
  - Research Site, Zuid-Scharwoude
  - Research Site, Zutphen